CLINICAL TRIAL: NCT03957525
Title: The Influence of a Pre-Operative Preparatory Virtual Reality Program on the Self-Assessed Anxiety of Children Undergoing Elective Surgery
Brief Title: Pediatric Preoperative Virtual Reality Program
Acronym: PPVRP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting process could not be completed; lack of participants
Sponsor: Thoralf Liebs (Other)
Responsible Party: Sponsor-Investigator, Thoralf Liebs, PD Dr. med. Thoralf R. Liebs, consultant orthopaedic surgeon, pediatric orthopaedics, special orthopedic surgery, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2019-00081
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Surgery; Anxiety
Keywords: Virtual reality; Pediatric; Anxiety; Surgery; Anesthesia; Intervention; Exposure; Randomized controlled trial; Pediatric urology; Orthopedic surgery; General Pediatric surgery; Pediatric orthopedics
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Prospective randomized, controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Orthopaedic Intervention group (Experimental): In addition to the written and oral preparation for surgery this arm receives an 'on-boarding' package containing a cardboard VR, a code to download the VR App and a plush penguin.
  Interventions: Other: Pre-Operative Preparatory Virtual Reality Program
- Orthopaedic Control group (No Intervention): Gets written and oral preparation for surgery
- Urologic Intervention group (Experimental): In addition to the written and oral preparation for surgery this arm receives an 'on-boarding' package containing a cardboard VR, a code to download the VR App and a plush penguin.
  Interventions: Other: Pre-Operative Preparatory Virtual Reality Program
- Urologic Control group (No Intervention): Gets written and oral preparation for surgery
- General Paediatric Surgery Intervention group (Experimental): In addition to the written and oral preparation for surgery this arm receives an 'on-boarding' package containing a cardboard VR, a code to download the VR App and a plush penguin.
  Interventions: Other: Pre-Operative Preparatory Virtual Reality Program
- General Paediatric Surgery Control group (No Intervention): Gets written and oral preparation for surgery

INTERVENTIONS:
Other: Pre-Operative Preparatory Virtual Reality Program — The Influence of a Pre-Operative Preparatory Virtual Reality Program on the Self-Assessed Anxiety of Children Undergoing Elective Surgery
  Arms: General Paediatric Surgery Intervention group; Orthopaedic Intervention group; Urologic Intervention group

SUMMARY:
Does the introduction of a preparatory virtual reality (VR) program that is used in the home environment, have an effect on the anxiety level of children immediately before surgery, prior to administration of preoperative sedatives?

DETAILED DESCRIPTION:
Up to 60% of children who require elective surgery report significant anxiety in the preoperative setting. Severe perioperative anxiety of a child poses a major challenge for the surgeon, since it is often accompanied by adverse behavioral and emotional reactions and associated with a complicated operative and postoperative course.

The investigators have made the personal experience that informing the children ahead of time about what to expect in the hospital, decreases child anxiety and increases parent satisfaction.

There is considerable debate on the best way how to inform children about what to expect during their hospital stay. The investigators had a virtual reality application developed that introduces the children to several aspects of the hospital environment. Therefore, these children now ahead of time what they will experience during their hospital stay.

The aim is to evaluate the effect of this preparatory virtual reality application on the anxiety level of children immediately before surgery.

ELIGIBILITY:
Inclusion Criteria:

1. The child is between the age of 7 and 13 years
2. The child is undergoing an elective surgical procedure under general anesthesia
3. The child understands Swiss German
4. The parent(s) understand(s) German
5. The parent(s) possess a smart phone
6. Internet access is given
7. The patient information has been explained
8. Informed Consent is signed

Exclusion Criteria:

1. The child has a hearing impairment
2. The child has neurologic disorder
3. The child requires postoperative intensive care
4. The child has previous experience of anesthesia
5. American Society of Anesthesiologists (ASA) score of III or greater

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Perioperative anxiety level of children immediately before surgery (VAS-A) | 2 - 90 days after recruiting
  Perioperative anxiety level of children as measured by the Visual Analog Scale for Anxiety (VAS-A), immediately before surgery, prior to administration of preoperative sedatives (T2).
  The VAS-A scale consists of a 10 cm long, horizontal line, supplemented by two labels: "no anxiety or fear" at the left end, "worst possible anxiety or fear" at the right end of the scale.

SECONDARY OUTCOMES:
Perioperative anxiety level of Children VAS-A | 2 - 90 days after recruiting
  Perioperative anxiety level of children measured at T0, T1 and T3 with VAS-A.
Perioperative anxiety level of Children VFAS | 2 - 90 days after recruiting
  Perioperative anxiety level of children as measured by the Visual Faces Analog Scale (VFAS) scale at T0, T1, T2 and T3.
  The VFAS scale consists of six different drawings of faces, supplemented by labels as follows: ("Anxiety Level:", "none", "mild", "mild-moderate", "moderate", "moderate-high", "highest")
Perioperative anxiety level of accompanying parent | 14 - 110 days after recruiting
  Perioperative anxiety level of accompanying parent measured at T0, T1 and T2 with the VAS-A and VFAS scale
Non-disease specific secondary Outcomes | 14 - 110 days after recruiting
  The investigators want to evaluate to which extent the VR program is able to improve the patient and parent's level of preparedness for surgery. Unfortunately, there are currently no validated outcome measures available covering these issues. Therefore, we developed a questionnaire assessing the level of preparedness related to seven aspects of the hospital stay, which are particularly illustrated by the VR program.

CONTACTS AND LOCATIONS:
Overall Officials: Thoralf Randolf Liebs, PD Dr. med, Principal Investigator — Department of Pediatric Surgery, Inselspital
Locations (1):
- Inselspital Bern, Clinic for Pediatric Surgery, Bern, Switzerland